CLINICAL TRIAL: NCT03186339
Title: Validation of the "Toronto Aortic Stenosis Quality of Life Questionnaire" in Patients Undergoing Surgical Aortic Valve Replacement or Transfemoral Transcatheter Aortic Valve Implantation The TASQ Registry
Brief Title: Validation of the "TASQ" in Patients Undergoing SAVR or TF-TAVI
Acronym: TASQ
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IPPM2017TASQ
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Aortic Valve Stenosis
Keywords: QoL; TAVI; surgical aortic valve replacement; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TAVI patients: patients undergoing TF (transfemoral) TAVI as treatment for the aortic stenosis
  Interventions: Procedure: TAVI
- SAVR patients: patients undergoing isolated surgical valve replacement as treatment for the aortic stenosis
  Interventions: Procedure: SAVR
- MM patients: patients in whom the aortic stenosis is medically managed
  Interventions: Other: MM

INTERVENTIONS:
Procedure: TAVI — transfemoral transcatheter aortic valve implantation
  Groups: TAVI patients
Procedure: SAVR — isolated surgical valve replacement
  Groups: SAVR patients
Other: MM — management of aortic stenosis by medical treatment only
  Groups: MM patients

SUMMARY:
Prospective, multi-centre, multi-national registry with a follow-up of 3 months, in five European countries and Canada (Toronto), with elective patients undergoing TF-TAVI (n=120) and isolated SAVR (n=120), respectively and a control group of 50 patients receiving medical treatment only. All patient groups will fill in three different questionnaires to assess quality of life in 5 different languages (English, French, German, Italian and Spanish). One of these will be a new questionnaire, the Toronto Aortic Stenosis QoL (Quality of Life) questionnaire (TASQ).

DETAILED DESCRIPTION:
Currently, there are two cardiovascular disease QoL scales which have been used in studies of patients with aortic stenosis - the Minnesota Living with Heart Failure (MLHF) questionnaire and the Kansas City Cardiomyopathy Questionnaire (KCCQ).

The KCCQ has now become the only cited health related (HR) QoL validated scale for use among a growing TAVI (Transcatheter Aortic Valve Implantation) patient population; however questions on the KCCQ do not reflect the concerns and lifestyle of patients proceeding for aortic valve intervention. Many of the questions do not reflect this patient population's perspective of well-being in contrast to perceptions by the general cardiac population on which it was validated. It is important to capture the disruptions caused by a chronic disease and its treatment on lifestyles, activities, and interests; that is interference with psychologically meaningful activity. It has been noted that this interference varies by disease process and treatment by general scales such as the Illness Intrusiveness Scale .

Due to issues of limited validity of the KCCQ for TAVI / SAVR (Surgical Aortic Valve Replacement) patients related to symptom items not being revised from their original use for congestive heart failure, a new original HR-QoL questionnaire was proposed: The "Toronto Aortic Stenosis Quality of Life Questionnaire" (TASQ) is a health specific measurement tool designed to measure changes in quality of life in aortic stenosis patients. The aim of this study is to validate this questionnaire in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* severe aortic stenosis
* age > 18 years
* in case of TAVI or SAVR: intention to treat the AS employing an Edwards valve

Exclusion Criteria:

* patients not providing informed consent
* patients with major cognitive impairment
* emergency patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 120 consecutive patients undergoing TF-TAVI, 120 patients undergoing SAVR, and a control group of 50 patients receiving medical treatment will be enrolled. Because of an expected loss during follow-up with not all patients returning this will result in about 100 patients for both TAVI and SAVR and 40 for medical management or 48 per language.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Change in QoL as assessed by SF12 (Short Form 12) Questionnaire | 3 months from baseline examination
  Change in quality of life as assessed by the SF12 using a points system
Change in QoL as assessed by KCCQ (The Kansas City Cardiomyopathy Questionnaire) | 3 months from baseline examination
  Change in quality of life as assessed by the KCCQ using a points system
Change in QoL as assessed by TASQ (Toronto Aortic Stenosis Quality of Life Questionnaire) | 3 months from baseline examination
  Change in quality of life as assessed by the TASQ using a points system

SECONDARY OUTCOMES:
Difference in change in QoL between arms | 3 months from baseline examination
  Difference in change in QoL between the three intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Rima Styra, MD, Principal Investigator — University Health Network, Toronto General Hospital, Ontario, Canada; Derk Frank, Prof., Principal Investigator — UKSH University Clinical Center Schleswig-Holstein, Germany; Simon Kennon, MD, Principal Investigator — Barts Heart Centre, London, UK
Locations (10):
- Medical University of Innsbruck, Innsbruck, Austria
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada
- France (2):
  - Hospital Jacques Cartier, Massy
  - Bichat Hospital - Claude-Bernard, Paris
- UKSH University Clinical Center Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany
- Italy (2):
  - Structual Interventional Cardiology, University Hospital Careggi, Florence
  - Department of Medicine, University of Verona, Verona
- Spain (2):
  - Hospital Juan Canalejo Coruna, A Coruña
  - University Hospital Vall d'Hebron, Barcelona
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frank D, Kennon S, Bonaros N, Romano M, Lefevre T, Di Mario C, Stefano P, Ribichini FL, Himbert D, Urena-Alcazar M, Salgado-Fernandez J, Cuenca Castillo JJ, Garcia B, Kurucova J, Thoenes M, Luske C, Bramlage P, Styra R. Trial protocol for the validation of the 'Toronto Aortic Stenosis Quality of Life (TASQ) Questionnaire' in patients undergoing surgical aortic valve replacement (SAVR) or transfemoral (TF) transcatheter aortic valve implantation (TAVI): the TASQ registry. Open Heart. 2019 May 21;6(1):e001008. doi: 10.1136/openhrt-2019-001008. eCollection 2019. PMID 31218003
- [Result] Frank D, Kennon S, Bonaros N, Stastny L, Romano M, Lefevre T, Di Mario C, Stefano P, Ribichini F, Himbert D, Urena-Alcazar M, Salgado-Fernandez J, Castillo JJC, Garcia Del Blanco B, Deutsch C, Sykorova L, Kurucova J, Thoenes M, Luske CM, Bramlage P, Styra R. Aortic valve replacement: validation of the Toronto Aortic Stenosis Quality of Life Questionnaire. ESC Heart Fail. 2021 Feb;8(1):270-279. doi: 10.1002/ehf2.12961. Epub 2020 Nov 18. PMID 33207035
- [Result] Kennon S, Styra R, Bonaros N, Stastny L, Romano M, Lefevre T, Di Mario C, Stefano P, Ribichini FL, Himbert D, Urena-Alcazar M, Salgado-Fernandez J, Cuenca Castillo JJ, Garcia B, Deutsch C, Sykorova L, Kurucova J, Thoenes M, Luske C, Bramlage P, Frank D. Quality of life after transcatheter or surgical aortic valve replacement using the Toronto Aortic Stenosis Quality of Life Questionnaire. Open Heart. 2021 Nov;8(2):e001821. doi: 10.1136/openhrt-2021-001821. PMID 34810276